CLINICAL TRIAL: NCT00624117
Title: Progressive Exercise After Operation of Rotator Cuff Rupture and Anterior Labrum Rupture: Randomized Controlled Trial
Brief Title: Progressive Exercise After Operation of Rotator Cuff Rupture and Anterior Labrum Rupture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jyväskylä Central Hospital (Other)
Responsible Party: Jari Ylinen, MD, PhD, Jyväskylä Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dnro46/2005
Record Dates: First submitted 2008-02-15; First posted 2008-02-26 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2010-05

CONDITIONS: Rotator Cuff Disease; Shoulder Joint
Keywords: shoulder joint; recovery of function; effectiveness of rehabilitation; rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Behavioral: Progressive exercise

INTERVENTIONS:
Behavioral: Progressive exercise — home-based exercise program, 2 to 3 exercise sessions per week

SUMMARY:
The purpose of this study is to evaluate the effectiveness of progressive strength training after rotator cuff and labrum operation of the shoulder joint.

ELIGIBILITY:
Inclusion Criteria:

* rupture of rotator cuff
* rupture of anterior labrum
* age 18 to 65 years
* motivated to continue in work life
* motivated for rehabilitation

Exclusion Criteria:

* former operation in the same joint
* major arthrosis in the same joint
* cervical disk herniation
* concised spinal cord
* conditions after cervical spine operations
* rheumatic diseases
* fibromyalgia
* pregnancy
* severe depression
* alcoholism
* misusing of drugs
* disease that prevents progressive exercise eg. back pain, heart disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-05; Primary Completion 2009-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Strength and mobility | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jari Ylinen, PhD, Principal Investigator — Jyväskylä Central Hospital
Locations (1):
- Jyväskylä Central Hospital, Jyväskylä, Finland